CLINICAL TRIAL: NCT02069730
Title: Genomic Profiling and Matched Therapy for Recurrent or Metastatic Salivary Gland Neoplasms
Brief Title: A Study of Drug Therapies for Salivary Gland Cancers Based on Testing of Genes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEMS-001
Record Dates: First submitted 2014-02-20; First posted 2014-02-24 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Salivary Gland Cancer; Metastatic; Advanced; Recurrent
Keywords: molecular profiling; selinexor; tumor tissue
MeSH Terms: conditions — Salivary Gland Neoplasms; Neoplasm Metastasis; Recurrence; Neoplasms | interventions — selinexor; Androgen Antagonists; Mitogen-Activated Protein Kinase Kinases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unmatched Treatment (Selinexor) (Experimental): Selinexor, 30mg/m2, by mouth, twice weekly, every 28 day cycles.
  If patients have a "druggable" aberration but there is no access to the relevant agent, then patients will receive selinexor
  Interventions: Drug: Selinexor
- Matched Therapy (Experimental): EGFR or HER2 Inhibitor,FGFR Inhibitor,C-KIT Inhibitor, Anti-androgen ,NOTCH Inhibitor,MEK or PI3K Inhibitor .
  If the matched therapy is given through a clinical trial, the dosing schedule will be determined by that particular trial protocol. For matched treatments administered outside of a clinical trial, the dosing schedule will be the recommended dose by the expertise of the treating investigator.
  Interventions: Drug: EGFR or HER2 Inhibitor; Drug: FGFR Inhibitor; Drug: C-KIT Inhibitor; Drug: Anti-androgen; Drug: NOTCH Inhibitor; Drug: MEK or PI3K Inhibitor

INTERVENTIONS:
Drug: Selinexor — If no "druggable" aberrations are identified on the molecular profiling analysis, then patients will receive unmatched treatment with Selinexor, a selective inhibitor of nuclear export (SINE).
  Other Names: KPT-330
  Arms: Unmatched Treatment (Selinexor)
Drug: EGFR or HER2 Inhibitor — If specific "druggable" aberrations are identified on the molecular profiling analysis, then patients will receive matched treatment with EGFR or HER2 Inhibitor
  Other Names: Matched treatment
  Arms: Matched Therapy
Drug: FGFR Inhibitor — If specific "druggable" aberrations are identified on the molecular profiling analysis, then patients will receive matched treatment with FGFR Inhibitor
  Other Names: Matched treatment
  Arms: Matched Therapy
Drug: C-KIT Inhibitor — If specific "druggable" aberrations are identified on the molecular profiling analysis, then patients will receive matched treatment with C-KIT Inhibitor
  Other Names: Matched Treatment
  Arms: Matched Therapy
Drug: Anti-androgen — If specific "druggable" aberrations are identified on the molecular profiling analysis, then patients will receive matched treatment with Anti-androgens
  Other Names: Matched Treatment
  Arms: Matched Therapy
Drug: NOTCH Inhibitor — If specific "druggable" aberrations are identified on the molecular profiling analysis, then patients will receive matched treatment with NOTCH Inhibitor
  Other Names: Matched Treatment
  Arms: Matched Therapy
Drug: MEK or PI3K Inhibitor — If specific "druggable" aberrations are identified on the molecular profiling analysis, then patients will receive matched treatment with MEK or PI3K Inhibitor
  Other Names: Matched Treatment
  Arms: Matched Therapy

SUMMARY:
This is a study of select drug therapies in patients with salivary gland cancer. The study has two phases: a molecular profiling phase (phase 1) and a treatment phase (phase 2).

Based on the Molecular profiling results in phase the participants will receive matched treatment if a specific aberration is identified or will receive treatment with Selinexor if unmatched and no druggable aberration is identified.

DETAILED DESCRIPTION:
In molecular profiling phase of the study, participants will provide a sample of their tumor tissue to test for changes in certain genes that show whether certain drug treatments will be more useful than others.

Once participants have undergone molecular profiling, they will be offered a drug treatment depending on the results. Certain drug treatments are designed to target certain gene changes. If there is a matching drug treatment, participants will be offered that treatment (either outside a clinical trial or within a clinical trial). If there are no gene changes or there are changes to genes were there are no drug treatments available for those certain changes, participants will be offered the study drug, Selinexor.

Cancer is the uncontrolled growth of cells. Research shows that one way cancer cells can grow uncontrollably is when certain proteins, called exporter proteins, are present in high levels in the body. These proteins prevent certain other proteins important in protecting cells from becoming cancerous and important in the controlling the growth of cells, from working. The study drug Selinexor is new class of drug called Selective Inhibitor of Nuclear Export (SINE) that blocks the exporter proteins from working which may allow the other proteins to work and slow or stop tumors from growing.

ELIGIBILITY:
Inclusion Criteria (Phase 1, Molecular Profiling):

* Have available archival tumor tissue or fresh tumor specimen from diagnostic histological tissue for molecular profiling.
* Histological or cytological proof of malignant salivary gland tumor
* ECOG performance score 0-2
* Documented evidence of recurrent or metastatic disease

Inclusion Criteria (Phase 2, Treatment):

* Interpretable result of molecular profiling in the molecular profiling phase of this study
* Advanced recurrent or metastatic salivary gland cancer for which no curative therapy exists
* Evidence of clinical or radiological disease progression at the time of study treatment
* At least one measurable target lesion as defined by RECIST 1.1
* Must have adequate hematological, liver, renal and cardiac function
* No concomitant use of drugs which may prolong QTc interval
* No history of serious cardiac illness
* No serious medical conditions that might be aggravated by treatment or limit compliance.
* Central nervous system metastases are permitted provided these are clinically stable
* Able to take oral medication and have no evidence of bowel obstruction, infectious/inflammatory bowel disease
* No other active malignancy at any other site
* 18 years of age or older
* Measureable disease as defined by RECIST v1.1
* Not receiving any other concurrent investigational agent
* If the matched treatment is in the context of another phase I trial, the eligibility criteria of the enrolled trial will be used instead of the criteria from this trial

Exclusion Criteria (Phase 1, Molecular Profiling):

* Refuses to have tumor tissue undergo molecular profiling
* Not enough tumor tissue for molecular profiling
* Life expectancy less than 3 months

Exclusion Criteria (Phase 2, Treatment):

* Had stopped the previous treatment but showed no clinical or radiological evidence of disease progression
* Have received the same drug treatment of assignment to the specific arm before the enrolment in to treatment phase (phase 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2023-06 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with complete and partial response to unmatched therapy Selinexor compared to matched therapies | 4 years
  Overall Response rate in the setting of matched and unmatched therapy.

SECONDARY OUTCOMES:
Number of participants with complete, partial and/or stable disease to unmatched therapy Selinexor compared to matched therapies | 4 years
  Disease control Rate in the setting of matched and unmatched therapy.
Length of time that participant's disease does not worsen | 6 months
  Progression free survival rate in the setting of matched and unmatched therapy.
Percentage of each molecular aberrations in metastatic salivary gland tumors | 4 years
  Molecular profiling results in malignant salivary gland tumor

CONTACTS AND LOCATIONS:
Overall Officials: Anna Spreafico, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada